CLINICAL TRIAL: NCT05220007
Title: Effect of Presbyopic Correction Lens on Humphrey Visual Field Testing in Patients With Multifocal Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Naris Kitnarong, Associate professor, Siriraj Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIOLVF001
Record Dates: First submitted 2021-12-27; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Glaucoma; Cataract Senile
Keywords: cataract; glaucoma; multifocal intraocular lens; presbyopia; cataract surgery
MeSH Terms: conditions — Glaucoma; Cataract; Presbyopia

STUDY DESIGN:
Intervention Model Description: Non-randomized, prospective comparative study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glaucomatous arm (Experimental): Mild stage glaucomatous patients age more than 18 years old, a history of uneventful phacoemulsification with MIOL implantation at least 1 month before participation, distant best-corrected visual acuity (BCVA) equal to or better than 20/30, near BCVA at least Jaeger 2.
  Interventions: Diagnostic Test: Humphrey visual field testing
- Non-glaucomatous arm (Active Comparator): Pseudophakic participants without glaucoma, age more than 18 years old, a history of uneventful phacoemulsification with MIOL implantation at least 1 month before participation, distant best-corrected visual acuity (BCVA) equal to or better than 20/30, near BCVA at least Jaeger 2.
  Interventions: Diagnostic Test: Humphrey visual field testing

INTERVENTIONS:
Diagnostic Test: Humphrey visual field testing — Perimetry was performed with the Humphrey Field Analyzer (Carl Zeiss Meditec Inc). Participants performed a 30-2 or a 24-2 Swedish Interactive Threshold Algorithm (SITA) standard test with stimulus size III, and standard Humphrey background luminance of 31.5 apostilbs. The participants were selected by simple random sampling to perform the HVF test with presbyopic collection lenses followed by without presbyopic collection lenses, or without presbyopic collection lenses followed by with presbyopic collection lenses. The power of presbyopic correction lens at the testing distance of 33 cm (the bowl radius) was auto-calculated according to the recommendation by the Humphrey Field Analyzer's manufacturer, depending on the current refractive error and the patient's age.

SUMMARY:
Purpose of this study was to evaluate the effect of presbyopic correction lens on Humphrey visual field (HVF) testing in patients with 2 models of multifocal intraocular lens (MIOL) both with and without glaucoma. All participants performed HVF testing with presbyopic collection lenses and without presbyopic collection lenses on the same occasion (5-10 minutes between the test). The mean deviation (MD) and pattern standard deviation (PSD) were compared between with and without presbyopic collection lenses, between glaucoma and non-glaucoma and between 2 models of MIOL.

DETAILED DESCRIPTION:
This was a prospective comparative study in patients who underwent uneventful phacoemulsification with MIOL implantation at the Department of Ophthalmology, Faculty of Medicine, Siriraj Hospital, Mahidol University between June 2009 to July 2012. The study protocol was approved by the Siriraj Institutional Review Board complied with all of the principles set forth in the Declaration of Helsinki (1964) and its subsequent amendments. (certificate of approval number Si 003/2010). The written informed consent was obtained from each participant prior to participation. Each patient received a comprehensive eye examination with slit-lamp biomicroscopy, distant and near visual acuity, and auto-refraction. The eligible participants performed HVF 24-2 or 30-2 on the enrollment day with and without presbyopic correction lens. The participants were randomized to perform HVF with presbyopic collection lenses followed by without presbyopic collection lenses or without presbyopic collection lenses followed by with presbyopic collection lenses by simple randomization. Data collection included demographic data, distant (logMar) and near (Jaeger reading chart) BCVA, and HVF test result including mean deviation (MD), pattern standard deviation (PSD), test duration (minute), fixation loss, false positive, and false negative.

Multifocal intraocular lens characteristics There were two types of aspheric diffractive MIOL included in the study: TECNIS ZM900 (Abbott Medical Optics Inc, Santa Ana, CA, USA) and AcrySof IQ ReSTOR SN6AD1 (Alcon Laboratories, Inc., Irvine, CA, USA). The TECNIS ZM900 is a silicone 3-piece aspheric diffractive lens. The power of the add is +4.00 D with a 50/50 distance/near light distribution. The AcrySof IQ ReSTOR SN6AD1is an acrylic single-piece aspheric diffractive lens. The power of the add is +3.00 D with a 65/35 light distribution.

ELIGIBILITY:
Inclusion Criteria:

* Glaucomatous and non-glaucomatous patients
* Age older than 18 years
* A history of uneventful phacoemulsification with MIOL implantation at least one month before participation
* Distant best-corrected visual acuity (BCVA) equal to or better than 20/30
* Near BCVA of at least Jaeger 2

Exclusion Criteria:

* The inability to perform reliable visual field testing (fixation loss, false positive or false negative more than 25%)
* A history of postoperative complications
* Moderate to advanced visual field defects (MD less than - 6 dB)
* Any other concurrent ocular diseases, except well-controlled glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Mean deviation | at 1 day after enrollment
  Mean deviation from Humphrey visual field testing
Pattern standard deviation | at 1 day after enrollment
  Pattern standard deviation from Humphrey visual field testing

SECONDARY OUTCOMES:
Fixation loss (percent) | at 1 day after enrollment
  Fixation loss from Humphrey visual field testing
False negative (percent) | at 1 day after enrollment
  False negative from Humphrey visual field testing
False positive (percent) | at 1 day after enrollment
  False positive from Humphrey visual field testing
Test duration (minutes0 | at 1 day after enrollment
  Test duration from Humphrey visual field testing

CONTACTS AND LOCATIONS:
Overall Officials: Naris Kitnarong, M.D., M.B.A., Principal Investigator — Mahidol University
Locations (1):
- Naris Kitnarong, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aychoua N, Junoy Montolio FG, Jansonius NM. Influence of multifocal intraocular lenses on standard automated perimetry test results. JAMA Ophthalmol. 2013 Apr;131(4):481-5. doi: 10.1001/jamaophthalmol.2013.2368. PMID 23430147
- [Result] Farid M, Chak G, Garg S, Steinert RF. Reduction in mean deviation values in automated perimetry in eyes with multifocal compared to monofocal intraocular lens implants. Am J Ophthalmol. 2014 Aug;158(2):227-231.e1. doi: 10.1016/j.ajo.2014.04.017. Epub 2014 Apr 29. PMID 24784872
- [Result] Yohannan J, Wang J, Brown J, Chauhan BC, Boland MV, Friedman DS, Ramulu PY. Evidence-based Criteria for Assessment of Visual Field Reliability. Ophthalmology. 2017 Nov;124(11):1612-1620. doi: 10.1016/j.ophtha.2017.04.035. Epub 2017 Jul 1. PMID 28676280
- [Result] Kumar BV, Phillips RP, Prasad S. Multifocal intraocular lenses in the setting of glaucoma. Curr Opin Ophthalmol. 2007 Feb;18(1):62-6. doi: 10.1097/ICU.0b013e328011d108. PMID 17159450